CLINICAL TRIAL: NCT01119313
Title: A Phase II, Single-center, Randomized, Controlled, Double-blind Study to Assess Effects on Skin Conditions and Patient Reported Outcome of a Topical Formulation Containing LAS41002 on Lesional Skin in Patients With Atopic Eczema
Brief Title: Study to Investigate Skin Conditions and Patient Assessment of LAS 41002 in the Treatment of Atopic Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: godehard.ocker, Almirall Hermal GmbH
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H 527 000-0917; 2009-017407-28 (EudraCT Number)
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAS 41002 (Experimental)
  Interventions: Drug: LAS 41002
- Active (Active Comparator)
  Interventions: Drug: Active

INTERVENTIONS:
Drug: LAS 41002 — LAS 41002, once daily
  Arms: LAS 41002
Drug: Active — Active, once daily
  Arms: Active

SUMMARY:
The aim of the study is an intra-individual comparison of skin conditions in addition to a patient based assessment of product appearance in the topical treatment of atopic eczema.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 years or older;
* two comparable treatment areas (difference in local SCORAD not greater than 3) on opposite extremities of 100 - 300 cm2 with at least one lesional region within each of these areas of ≥ 20 cm². Clinical condition of atopic eczema mild to moderate defined by a local SCORAD of at least 5 with

  1. erythema ≥ 2
  2. lichenification ≥ 1
  3. dryness ≥ 1
  4. itching ≥ 1
* Erlangen atopy score sum equal or higher than 10 points (3);
* the physical examination must be without disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the study;
* female patients of childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1 % per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices [IUDs], sexual abstinence or vasectomized partner;
* written informed consent obtained

Exclusion Criteria:

* acne, suntan, eczema, hyperpigmentation or tattoos in the test areas;
* dark-skinned persons whose skin color prevents ready assessment of skin reactions;
* evidence of drug or alcohol abuse;
* pregnancy or nursing;
* UV-therapy within 6 weeks before first treatment;
* symptoms of a clinically significant illness that may influence the outcome of the study in the four weeks before and during the study;
* participation in the treatment phase of another clinical study within the last four weeks prior to the first administration of investigational drug in this study;
* known allergic reactions to components of the study preparations, hypersensitivity against cetostearyl alcohol;
* treatment with systemic or locally acting medications which might counter or influence the study aim (e.g. antihistamines or glucocorticosteroids) within two weeks before study day 1and throughout the study period (exception: asthma may be found in patients with atopic eczema, therefore inhalation with corticosteroids in patients with asthma accompanying atopic eczema will be allowed at a dose not exceeding 1 mg/day. The dosage should remain constant throughout the study period);
* contraindications according to summary of product characteristics;
* in the opinion of the investigator or physician performing the initial examination the patient should not participate in the study, e.g. due to probable noncompliance or inability to understand the study and give adequately informed consent;
* patient is institutionalized because of legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in total sum score of Clinical signs | 15 days
  scoring of clinical parameters (erythema, edema, crusting, excoriation, lichenification, dryness, itching) will be performed on a 4 point scale by investigator, comparing data from baseline (day1) vs end of trial (day15)

SECONDARY OUTCOMES:
change in skin hydration | 15 days
  measurement will be performed by corneometry, comparing data from baseline (day1) vs end of trial (day15)
Time dependancy of Skin penetration | 2 hours
  subject's 5 point assessment of perceived skin penetration will be performed for 2 hours after the first application
patient overall assessment | 15 days
  patient's intraindividual 5 point assessment on product on perception will be performed at end of trial (day15)
Number of skin reactions per patient as a measure of safety and tolerability | 15 days
  scoring will be performed by investigator
Number of Adverse Events per patients as a measure of safety and tolerability | Daily
  reporting will be performed by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (1):
- Almirall Investigational Sites#1, Hamburg, Germany

REFERENCES:
- [Derived] Ruzicka T, Willers C, Wigger-Alberti W. Efficacy and patient-reported outcomes of a new mometasone cream treating atopic eczema. Skin Pharmacol Physiol. 2012;25(6):305-12. doi: 10.1159/000341809. Epub 2012 Aug 31. PMID 22948032
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp